CLINICAL TRIAL: NCT07351864
Title: Impact of Finerenone in Combination With Sodium Glucose Cotransporter-2 Inhibitor in Patients With Heart Failure
Brief Title: Finerenone Plus SGLT2 Inhibitors in Heart Failure
Acronym: FIN-SGLT2-HF
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mansour Saad, PhD Candidate in Clinical Pharmacy, Mansoura University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MDP.25.08.190
Record Dates: First submitted 2025-12-28; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Heart Failure
Keywords: Finerenone; SGLT2 inhibitor; Dapagliflozin; Heart failure therapy; Cardioprotection
MeSH Terms: conditions — Heart Failure | interventions — finerenone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Finerenone Plus SGLT-2 inhibitor (dapagliflozin) (Experimental): Participants in this arm will receive finerenone in addition to standard therapy with a sodium-glucose cotransporter-2 (SGLT2) inhibitor (dapagliflozin). Finerenone will be administered at a dose of 10 mg once daily and dapagliflozin will be administered at a dose of 10 mg once daily, according to standard clinical practice
  Interventions: Drug: Finerenone; Drug: dapagliflozine
- SGLT-2 inhibitor (dapagliflozin) alone (Active Comparator): Participants in this arm will receive standard therapy with a sodium-glucose cotransporter-2 (SGLT2) inhibitor (dapagliflozin) alone. Dapagliflozin will be administered at a dose of 10 mg once daily according to standard clinical practice.
  Interventions: Drug: dapagliflozine

INTERVENTIONS:
Drug: Finerenone — Finerenone administered orally at a dose of 10 mg once daily.
  Arms: Finerenone Plus SGLT-2 inhibitor (dapagliflozin)
Drug: dapagliflozine — Dapagliflozin administered orally at a dose of 10 mg once daily.

SUMMARY:
The goal of this clinical study is to evaluate whether adding finerenone to standard treatment with a sodium-glucose cotransporter-2 (SGLT2) inhibitor provides additional benefits in patients with heart failure.

The main question this study aims to answer is whether the combination of finerenone and an SGLT2 inhibitor improves clinical outcomes and is safe compared to treatment with an SGLT2 inhibitor alone.

Participants will receive standard therapy with an SGLT2 inhibitor, with or without the addition of finerenone and will be followed to assess clinical outcomes and safety.

DETAILED DESCRIPTION:
Heart failure is a chronic clinical syndrome associated with significant morbidity, mortality and healthcare burden worldwide, despite advances in pharmacological therapy. Sodium-glucose cotransporter-2 (SGLT2) inhibitors have become an important component of standard treatment for patients with heart failure due to their demonstrated cardiovascular benefits. However, a substantial residual cardiovascular risk persists, indicating the need for additional therapeutic strategies.

Finerenone is a nonsteroidal mineralocorticoid receptor antagonist with a distinct mechanism of action that targets mineralocorticoid receptor activation in cardiac and renal tissues. Previous clinical studies have demonstrated that finerenone reduces inflammation and fibrosis and provides cardiovascular benefits in patients with chronic cardiovascular and renal diseases. These findings support the potential for finerenone to offer complementary cardioprotective effects when combined with established heart failure therapies.

This prospective controlled pilot study is designed to evaluate the clinical effects and safety of adding finerenone to standard therapy with an SGLT2 inhibitor in patients with heart failure, compared with treatment using an SGLT2 inhibitor alone. Patients receiving stable SGLT2 inhibitor therapy will be managed according to the assigned treatment strategy and followed throughout the study period to evaluate overall clinical outcomes and safety parameters.

The findings of this pilot study are expected to provide preliminary evidence regarding the potential benefits and tolerability of combining finerenone with SGLT2 inhibitors in patients with heart failure and to inform the design of future larger-scale clinical studies.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged 18 - 65 years.
* Newly diagnosed with HFrEF or HFpEF.
* Clinically stable and eligible to start SGLT2 inhibitors ± Finerenone therapy.

Exclusion Criteria:

* Patients with stroke.
* eGFR <25 mL/min.
* HF secondary to congenital heart disease or pulmonary hypertension
* Use intravenous inotropes.
* Patients needing cardiac transplantation.
* Known allergy to study medications.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-18 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular Mortality and Heart Failure Hospitalization | Up to 12 weeks (assessed at Baseline, Week 4, and Week 12)
  Incidence of cardiovascular mortality and hospitalization due to heart failure in each treatment group.

SECONDARY OUTCOMES:
All-cause Mortality | Up to 12 weeks (assessed at Baseline, Week 4, and Week 12)
  Number of participants with all-cause mortality in each treatment group.
Change in NYHA Functional Class | Up to 12 weeks (assessed at Baseline, Week 4, and Week 12)
  Change in New York Heart Association (NYHA) functional class in each treatment group.
Change in Serum Potassium Level | Up to 12 weeks (assessed at Baseline, Week 4, and Week 12)
  Serum potassium concentration (mmol/L) measured at baseline, Week 4 and Week 12 in each treatment group.
Change in Estimated Glomerular Filtration Rate (eGFR) | Up to 12 weeks (assessed at Baseline, Week 4, and Week 12)
  Estimated glomerular filtration rate (eGFR, mL/min/1.73 m²) measured at baseline, Week 4 and Week 12 in each treatment group.
Change in Kansas City Cardiomyopathy Questionnaire (KCCQ) Overall Summary Score | Baseline and Week 12
  Change in health-related quality of life assessed using the Kansas City Cardiomyopathy Questionnaire (KCCQ) overall summary score in each treatment group. Scores range from 0 to 100, with higher scores indicating better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Mansour Saad Alqahtani, PhD Candidate, Principal Investigator — Faculty of pharmacy, Mansoura university
Locations (1):
- Mansoura University Hospitals, Cardiology Department (Specialized Medical Hospital), Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared outside the study team as the study is conducted for academic research purposes and data confidentiality will be maintained.

REFERENCES:
- [Result] Filippatos G, Anker SD, Agarwal R, Ruilope LM, Rossing P, Bakris GL, Tasto C, Joseph A, Kolkhof P, Lage A, Pitt B; FIGARO-DKD Investigators. Finerenone Reduces Risk of Incident Heart Failure in Patients With Chronic Kidney Disease and Type 2 Diabetes: Analyses From the FIGARO-DKD Trial. Circulation. 2022 Feb 8;145(6):437-447. doi: 10.1161/CIRCULATIONAHA.121.057983. Epub 2021 Nov 13. PMID 34775784
- [Result] Pamporis K, Karakasis P, Sagris M, Zarifis I, Bougioukas KI, Pagkalidou E, Milaras N, Samaras A, Theofilis P, Fragakis N, Tousoulis D, Xanthos T, Giannakoulas G. Mineralocorticoid receptor antagonists in heart failure with reduced ejection fraction: a systematic review and network meta-analysis of 32 randomized trials. Curr Probl Cardiol. 2024 Jul;49(7):102615. doi: 10.1016/j.cpcardiol.2024.102615. Epub 2024 Apr 29. PMID 38692445
- [Result] Bakris GL, Agarwal R, Anker SD, Pitt B, Ruilope LM, Rossing P, Kolkhof P, Nowack C, Schloemer P, Joseph A, Filippatos G; FIDELIO-DKD Investigators. Effect of Finerenone on Chronic Kidney Disease Outcomes in Type 2 Diabetes. N Engl J Med. 2020 Dec 3;383(23):2219-2229. doi: 10.1056/NEJMoa2025845. Epub 2020 Oct 23. PMID 33264825